CLINICAL TRIAL: NCT05045768
Title: Treatment of Postinfectious Irritable Bowel Syndrome and Noninfective Irritable Bowel Syndrome With Gelsectan
Brief Title: Postinfectious Irritable Bowel Syndrome and Gelsectan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Consultant Gastroenterologist, Evangelismos Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 348/28-7-2021
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; postinfectious; xyloglycan
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postinfectious ibs and diarrhea predominant classical IBS (Experimental): Capsule containing Tamarind seed polysaccharide containing xyloglucan, combined with a pea protein reticulated with grape seed extractand a prebiotic, the xilooligosaccharide (Gelsectan, Devintec sagl) twice daily
  Interventions: Drug: (Gelsectan, Devintec Sagl)

INTERVENTIONS:
Drug: (Gelsectan, Devintec Sagl) — Patients included in the study will receive for 28 days a capsule containing Xyloglucan, Pea Protein and Grape Seed Extract and a prebiotic Xylo-oligosaccharide (Gelsectan, Devintec sagl) twice daily.

SUMMARY:
Irritable Bowel Syndrome (IBS) is one of the most common conditions diagnosed in gastroenterology practice. Acute infectious gastroenteritis represents the strongest known risk factor for IBS development; a condition known as post-infection IBS (PI-IBS). PI-IBS patients are more likely than sporadic IBS patients to exhibit a diarrhea-predominant phenotype. The investigators plan to prospectively recruit two groups of patients: patients with diarrhea-predominant post-infectious IBSand patients with diarrhea predominant classical IBS (non PI-IBS) who will be used as controls.

Patients included in the study will receive for 28 days a capsule containing Tamarind seed polysaccharide containing xyloglucan, combined with a pea protein reticulated with grape seed extractand a prebiotic, the xilooligosaccharide (Gelsectan, Devintec Sagl) twice daily.

DETAILED DESCRIPTION:
The Irritable bowel syndrome (IBS) is a functional disorder of alimentary system, which is recently considered as an erroneous gut-brain interaction. IBS is one of the most common conditions diagnosed in gastroenterology practice. Its prevalence ranges between 7-16% in western countries and is more common in females and younger individuals. Although the etiology of IBS is still obscure, its pathophysiology is dominated by a combination of both psychological factors and gastrointestinal dysfunction. Recent efforts have allowed identification of several peripheral micro-organic abnormalities. These include changes in gut microbiota, low grade mucosal inflammation, and epithelial dysfunction. Acute infectious gastroenteritis represents the strongest known risk factor for IBS development; a condition known as post-infectiousIBS (PI-IBS). According to a recent survey PI-IBS accounts for around 13% of all IBS. Today the diagnostic criteria for PI-IBS proposed by the Rome Foundation Working Team are based on the Rome IV criteria. These criteria were not part of the original Rome IV document as they were prepared after the release of Rome IV publications and need to be fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis. The acute infectious gastroenteritis is ideally diagnosed by stool culture (although only occasionally obtained in community subjects), validated molecular biology analyses (e.g., polymerase chain reaction) or by the presence of ≥2 of the following: fever, vomiting, or diarrhea. The investigators plan to prospectively recruit two groups of patients: patients with diarrhea-predominant post-infectious IBSand patients with diarrhea predominant classical IBS (non PI-IBS) who will be used as controls. Patients included in the study will receive for 28 days a capsule containing Xyloglucan, Pea Protein and Grape Seed Extract and a prebiotic Xylo-oligosaccharides (Gelsectan, Devintec sagl) twice daily. Drugs that might have any effect on intestinal motility or secretion will not be allowed during the study period.

Patients responding to treatment will be those in whom diarrhea disappeared, i.e. reported two or less non-watery stools emissions per day (stool of type 5 or less on the Bristol scale). Response to treatment will be assessed in the two group of patients immediately after the end of the 28-day administration of Gelsectan; however all patients will be followed for another 3 months and long term response to treatment will be assessed in that time period as well. The presence and intensity of abdominal pain and flatulence will also be measured on a seven-point Likert scale (7 very much better, 6 much better, 5 somewhat better, 4 same, 3 somewhat worse, 2 much worse, 1 very much worse). These measurements will be made in all patients immediately at the end of the 28-day administration of Gelsectan and at the end of the 3 month follow up period as well. Treatment response will be compared between the two groups using the chi squared test.

Safety and tolerability will be monitored during the entire study period through adverse events occurence.

ELIGIBILITY:
Inclusion Criteria:

Patients with diarrhea-predominant post-infectious IBSand patients with diarrhea predominant classical IBS (non PI-IBS) who will be used as controls

Diagnosis of IBS will be made according to the ROME iV criteria as following:

Recurrent abdominal pain, on average, at least 1 day/week in the last 3 months, associated with two or more of the following criteria:

* Related to defecation
* Associated with a change in frequency of stool
* Associated with a change in form (appearance) of stool. The above-mentioned criteria have to be fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.

Diagnosis of post infectious IBS will be made according to the Rome Foundation Working Team criteria as following:

Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, with symptom onset at least 6 months before diagnosis, associated with two of the following:

1. defecation
2. a change in frequency of stool
3. a change in form (appearance) of stool Symptom development immediately after resolution of acute infectious gastroenteritis

Infectious gastroenteritis should be defined by positive stool culture in a symptomatic individual or presence of two of the following acute symptoms (when stool culture not available):

1. fever
2. vomiting
3. diarrhea

Exclusion Criteria:

* Patients should not meet criteria for IBS before onset of acute illness.
* We will exclude patients who are pregnant, who have an oncology history (since these patients might exhibit diarrhea due to their underlying illness) and patients with alcohol dependence (due to the non-compliance shown by these patients) and patients with known hypersensitivity or allergy to any of the ingredients included in Gelsectan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Disappearance of diarrhea | After the end of the 28-day administration of xyloglycan
  Two or less non-watery stools emissions per day (stool of type 5 or less on the Bristol scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece